CLINICAL TRIAL: NCT03084783
Title: Dexamethasone in Herpes Simplex Virus Encephalitis Open Label Randomized Controlled Trial With an Observer-blinded Evaluation at 6 Months
Brief Title: Dexamethasone in Herpes Simplex Virus Encephalitis
Acronym: DexEnceph
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC16.015
Record Dates: First submitted 2017-02-03; First posted 2017-03-21 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: HSV Encephalitis
Keywords: dexamethasone; HSV encephalitis
MeSH Terms: conditions — Encephalitis, Herpes Simplex | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive dexamethasone 10mg intravenously 6 hourly for 4 days.
  Interventions: Drug: Dexamethasone
- Control group (No Intervention): Participants receive standard care and no dexamethasone.

INTERVENTIONS:
Drug: Dexamethasone — Participants receive dexamethasone 10mg intravenously 6 hourly for 4 days.
  Arms: Intervention group

SUMMARY:
Encephalitics is a serious condition in which the brain becomes inflamed (swollen). It usually happens as a direct result of virus, such as herpes simplex virus (HSV).

HSV encephalitis is often treated with the drug acyclovir (an antiviral drug which slows the growth and spread of HSV in the body). Despite this however, around 2 out of every 3 people will have memory difficulties long term. Dexamethasone is a corticosteroid medication, which works by preventing the release of natural chemicals in the body which cause inflammation. It is possible that dexamethasone could help to reduce in swelling of the brain may improve the recovery of patients with HSV encephalitis. The aim of this study is to find out whether treatment with dexamethasone can improve long-term health outcomes in adults with HSV Encephalitis.

ELIGIBILITY:
Inclusion Criteria:

- Suspected encephalitis criteria: Acute or subacute (up to 4 weeks) alteration in consciousness, cognition, personality or behaviour* persisting for > 24 hours Laboratory confirmed HSV by positive PCR on CSF sample.

* Receiving intravenous aciclovir dosed at 10mg/kg TDS or at a reduced dose in renal impairment
* Age ≥ 18 years
* Person affiliated to social security
* Written informed consent has been given by the patient or their legal representative

Exclusion Criteria:

* Currently receiving oral or injectable corticosteroid therapy; including treatment with oral or injectable corticosteroids in the last 30 days.
* History of hypersensitivity to corticosteroids
* Immunosuppression secondary to:

  * Known HIV infection & CD4 count under 200cell/mm3
  * Biologic therapy or other immunosuppressive agents [azathioprine, methotrexate, ciclosporin]
  * Solid organ transplant on immunosuppression
  * Bone marrow transplant
  * Currently undergoing a course of chemotherapy or radiotherapy
  * Known immunodeficiency syndrome [other than HIV]
  * Known haematological malignancy
* Pre-existing indwelling ventricular devices
* Peptic ulcer disease in the last 6 months: defined as a peptic ulcer seen at previous endoscopy or an upper gastrointestinal bleed causing ≥ 2 unit haemoglobin drop
* Currently on an antiretroviral regime containing rilpivirine
* Patients under legal protection, administrative or judicial control
* Pregnancy / Breast feeding and parturient
* Subject in exclusion period of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Calcul of verbal memory score | at 6 months post randomization
  The primary outcome is a verbal memory score as determined by the Wechsler Memory Scale (WMS-IV) Auditory Memory Index, at 6 months post randomisation.

SECONDARY OUTCOMES:
Visual Memory Index assessed by the Wechsler Memory Scale | 6 months and 18 months post randomization
  Neuropsychological outcome
Processing Working Memory - assessed by the Wechsler Adult Intelligence Scale version IV | 6 months and 18 months post randomization
  Neuropsychological outcome
Higher executive function -assessed by Trail Making Test Parts A and B | 6 months and 18 months post randomization
  Neuropsychological outcome
Anxiety -assessed by self-completed Beck Anxiety Inventory | 6 months and 18 months post randomization
  Neuropsychological outcome
Depression -assessed by self-completed Beck Depression Inventory Inventory | 6 months and 18 months post randomization
  Neuropsychological outcome
Cognitive Assessment assessed by Addenbrooke's Cognitive Assessment revised (ACE-III) | at 30 days/discharge, 6 and 18 months
Requirement of intensive care or high dependency admission | during 18 months
  clinical outcome
Time to recovery of Glasgow Coma Scale (GCS) | during 18 months
  clinical outcome
Incidence of epilepsy | during 18 months
  clinical outcome
Measurement of temporal lobe volume (as % of intra-cranial volume) | Baseline, 2 weeks, 6 months and 18 months
  Imaging Outcomes
Measurement of Whole brain volume (as % of intra-cranial volume) | Baseline, 2 weeks, 6 months and 18 months
  Imaging Outcomes
Transcriptomic and proteomic profiling on CSF | at baseline and 2 weeks
  Biomarker outcomes
Transcriptomic and proteomic profiling on blood | at baseline, 4 days, 2 weeks, and 6 months
  Biomarker outcome
Anti NMDA receptor antibody testing | at 6 months
  Biomarker outcome
Proportion of patients with detectable HSV in CSF | at 2 weeks
  Safety Outcome
Health Status Measured by the EuroQOL-5D-5L questionnaire | at 6 and 18 months
Quality of Life measured by SF-36 questionnaires | at 6 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul STAHL, Principal Investigator — University Hospital, Grenoble
Locations (8):
- France (8):
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Hôtel-Dieu, Nantes
  - Hôpital Bichat-Claude Bernard, APHP, Paris
  - CHU Rennes, Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Delafontaine, Saint-Denis
  - CHU Strasbourg, Strasbourg
  - CHRU de Nancy, Hopitaux de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitley RJ. Herpes simplex encephalitis: adolescents and adults. Antiviral Res. 2006 Sep;71(2-3):141-8. doi: 10.1016/j.antiviral.2006.04.002. Epub 2006 Apr 25. PMID 16675036
- [Background] Granerod J, Ambrose HE, Davies NW, Clewley JP, Walsh AL, Morgan D, Cunningham R, Zuckerman M, Mutton KJ, Solomon T, Ward KN, Lunn MP, Irani SR, Vincent A, Brown DW, Crowcroft NS; UK Health Protection Agency (HPA) Aetiology of Encephalitis Study Group. Causes of encephalitis and differences in their clinical presentations in England: a multicentre, population-based prospective study. Lancet Infect Dis. 2010 Dec;10(12):835-44. doi: 10.1016/S1473-3099(10)70222-X. Epub 2010 Oct 15. PMID 20952256
- [Background] Tunkel AR, Glaser CA, Bloch KC, Sejvar JJ, Marra CM, Roos KL, Hartman BJ, Kaplan SL, Scheld WM, Whitley RJ; Infectious Diseases Society of America. The management of encephalitis: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2008 Aug 1;47(3):303-27. doi: 10.1086/589747. PMID 18582201